CLINICAL TRIAL: NCT03500692
Title: MitraClip NT System Post -Marketing Surveillance Study
Brief Title: MitraClip NT System Post-marketing Surveillance Study - Japan
Acronym: MitraClip NT
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: 17-519
Record Dates: First submitted 2018-03-30; First posted 2018-04-18 (Actual); Results first posted 2021-04-15 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-06

CONDITIONS: Mitral Regurgitation; Mitral Valve Regurgitation
Keywords: Mitral Valve Regurgitation; MitraClip; MitraClip NT; Japan MitraClip NT Postmarketing Surveillance
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: Yes

GROUPS / COHORTS (1):
- MitraClip NT System: Percutaneous mitral valve repair using MitraClip NT System
  Interventions: Device: MitraClip NT System

INTERVENTIONS:
Device: MitraClip NT System — Percutaneous mitral valve repair using MitraClip NT System

SUMMARY:
The purpose of the MitraClip post-marketing clinical use surveillance study is to observe the frequency, type and degree of adverse device effects and adverse events in order to assure the safety of the new medical device, and to collect safety and efficacy information for evaluating the results of the clinical use.

DETAILED DESCRIPTION:
This study is a prospective, mutli-center, single-arm post-marketing clinical use surveillance study. The Surveillance will consecutively register patients with moderate to severe and severe mitral regurgitation (3+ and 4+ MR) in whom a MitraClip implant was attempted. Patients registered in the AVJ-514 clinical trial who received additional MitraClip procedures will be excluded from the Surveillance.

Patients will be evaluated at Baseline, Procedure, Discharge, 30 days, 1 year, 2 years and 3 years in Japanese medical centers.

ELIGIBILITY:
Inclusion Criteria: Refer to MitraClip IFU

Exclusion Criteria: Refer to MitraClip IFU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-marketing Surveillance will consecutively register patients with moderate to severe and severe mitral regurgitation (3+ and 4+ MR) in whom a MitraClip implant was attempted.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2022-03-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (40):
- Japan (40):
  - Nagoya Heart Center, Nagoya, Aichi-ken
  - Toyohashi Heart Center, Toyohashi, Aichi-ken
  - New Tokyo Hospital, Matsudo, Chiba
  - Tokyo Bay Urayasu Ichikawa Medical Center, Urayasu, Chiba
  - Ehime Prefectural Central Hospital, Matsuyama, Ehime
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Asahikawa Medical University Hospital, Asahikawa, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo Prefectural Amagasaki General Medical Center, Amagasaki, Hyōgo
  - Hyogo Brain and Heart Center, Himeji, Hyōgo
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Iwate Medical University Hospital, Morioka, Iwate
  - Tokai University Hospital, Isehara, Kanagawa
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - St. Marianna Medical University Hospital, Kawasaki, Kanagawa
  - Saiseikai Yokohamashi Tobu Hospital, Yokohama, Kanagawa
  - Saiseikai Kumamoto Hospital, Kumamoto, Kumamoto
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Miyazaki Medical Association Hospital, Miyazaki, Miyazaki
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - The Sakakibara Heart Institute of Okayama, Okayama, Okayama-ken
  - Kishiwada Tokushukai Hospital, Kishiwada, Osaka
  - Osaka City University Hospital, Osaka, Osaka
  - Osaka General Medical Center, Osaka, Osaka
  - Osaka University Hospital, Suita-shi, Osaka
  - National Cerebral and Cardiovascular Center, Suita-shi, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Shizuoka General Hospital, Shizuoka, Shizuoka
  - Juntendo University Hospital, Bunkyo, Tokyo
  - The University of Tokyo Hospital, Bunkyo, Tokyo
  - Mitsui Memorial Hospital, Chiyoda City, Tokyo
  - Sakakibara Heart Institute, Fuchū, Tokyo
  - Keio University Hospital, Shinjuku-Ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-Ku, Tokyo
  - Teikyo University Hospital, tabashi City, Tokyo
  - Tottori University Hospital, Yonago, Tottori
  - Toyama University Hospital, Toyama, Toyama
  - Tokushima Red Cross Hospital, Tokushima

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 500 subjects were enrolled at 40 sites April 2, 2018 to March 31, 2020.
Period: Overall Study
Arm/Group | MitraClip NT System
Started | 500
Completed (3 - year visit complete) | 259
Not Completed | 241
Not completed — Death | 163
Not completed — Lost to Follow-up | 75
Not completed — Termination Reasons | 3

BASELINE CHARACTERISTICS:
Arm/Group | MitraClip NT System
Number analyzed (Participants) | 500
Age, Continuous [Mean (Standard Deviation); unit: Years] | 77.92 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206
  Male | 294
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 500
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Japan | 500
Height [Mean (Standard Deviation); unit: Centimeters] | 156.96 (10.02)
Weight [Mean (Standard Deviation); unit: Kilograms] | 52.05 (10.68)
Body Mass Index [Mean (Standard Deviation); unit: Kg/m^2] | 21.01 (3.22)
Society of Thoracic Surgeons (STS) Score [Mean (Standard Deviation); unit: Percentage of Expected Mortality] — The STS score is a validated risk-prediction model for open surgery based on data from the STS National Adult Cardiac Surgery Database. In general, an STS predicted risk of surgical mortality of 4%-8% is considered intermediate risk and 8% or greater is considered high risk. As of November 15, 2018, The Society of Thoracic Surgeons released an updated short-term risk calculator to reflect the latest 2018 adult cardiac surgery risk models. The STS Calculator allows you to calculate a patient's risk of mortality and morbidities for the most commonly performed cardiac surgeries.
  Percentage of Expected Mortality | 11.95 (9.66)
Cardiovascular History [Count of Participants; unit: Participants] — Population: All available data has been presented.
  Participants
    Dyslipidemia: number analyzed (Participants) | 498
    Dyslipidemia | 216
    Hypertension | 300
    Prior Transient Ischemic Attack (TIA): number analyzed (Participants) | 492
    Prior Transient Ischemic Attack (TIA) | 13
    Prior Cerebrovascular Accident (CVA): number analyzed (Participants) | 496
    Prior Cerebrovascular Accident (CVA) | 89
    Prior Myocardial Infarction: number analyzed (Participants) | 494
    Prior Myocardial Infarction | 124
    Cardiac Arrhythmia: number analyzed (Participants) | 495
    Cardiac Arrhythmia | 358
    Atrial Fibrillation: number analyzed (Participants) | 357
    Atrial Fibrillation | 316
Cardiac Intervention History [Count of Participants; unit: Participants] — Population: All available data has been reported.
  Participants
    Prior Cardiac Surgeries | 89
    Percutaneous Coronary Interventions: number analyzed (Participants) | 493
    Percutaneous Coronary Interventions | 142
    CRT/CRT-D: number analyzed (Participants) | 497
    CRT/CRT-D | 86
Co-Morbidity [Count of Participants; unit: Participants] — Population: All available data has been reported
  Participants
    Currently Smoking: number analyzed (Participants) | 492
    Currently Smoking | 30
    Diabetes: number analyzed (Participants) | 498
    Diabetes | 144
    Renal Failure: number analyzed (Participants) | 497
    Renal Failure | 244
    Chronic Lung Diesase: number analyzed (Participants) | 489
    Chronic Lung Diesase | 77
    Peripheral Artery Disease: number analyzed (Participants) | 494
    Peripheral Artery Disease | 56
    Prior Major Bleeding: number analyzed (Participants) | 494
    Prior Major Bleeding | 13
    Cirrhosis: number analyzed (Participants) | 497
    Cirrhosis | 6
    Cancer: number analyzed (Participants) | 498
    Cancer | 66
Heart Valve Intervention [Count of Participants; unit: Participants] | 28
Prior Heart Failure Hospitalization Within 1 year [Count of Participants; unit: Participants] — Population: All available data has been reported.
  Participants
    number analyzed (Participants) | 499
    (all) | 321
Baseline Etiology of Mitral Regurgitation [Count of Participants; unit: Participants]
  Degenerative MR Only | 126
  Functional MR Only | 358
  Mixed | 16
Baseline Effective Regurgitant Orifice Area [Mean (Standard Deviation); unit: cm^2] — Effective regurgitant orifice area is an important and clinically significant index of regurgitation severity. Effective regurgitant orifice area is calculated by Doppler echocardiography as the ratio of regurgitant volume/regurgitant jet time-velocity integral. Population: Data was not available for all the subjects.
  cm^2
    number analyzed (Participants) | 460
    (all) | 0.40 (0.26)
Regurgitant Volume [Mean (Standard Deviation); unit: mL/beat] — Regurgitant volume as determined by the Echocardiographic Core Laboratory (ECL). In the presence of regurgitation of one valve, without any intracardiac shunt, the flow through the affected valve is larger than through other competent valves. The difference between the two represents the regurgitant volume. Population: Data was not available for all the subjects.
  mL/beat
    number analyzed (Participants) | 461
    (all) | 58.04 (27.61)
Left Ventricular Ejection Fraction (LVEF) [Mean (Standard Deviation); unit: Percentage Of Ejection Fraction] — Population: All available data has been reported.
  Percentage Of Ejection Fraction
    number analyzed (Participants) | 499
    (all) | 46.10 (14.93)
Left Ventricular End Systolic Volume (LVESV) [Mean (Standard Deviation); unit: mL] — Left Ventricular End Systolic Volume (LVESV) as measured by the Echocardiography Core Laboratory (ECL). Left Ventricular end-systolic volume (LVESV) measured using 2-dimensional echocardiography. The endocardium is traced at end-systole (frame prior to mitral valve opening or the minimum cavity area) in the 2- and 4-chamber views to calculate volumes. Population: All available data has been reported.
  mL
    number analyzed (Participants) | 458
    (all) | 93.54 (64.43)
Left Ventricular End Diastolic Volume (LVEDV) [Mean (Standard Deviation); unit: mL] — Left Ventricular End Diastolic Volume (LVEDV) as measured by the site. Left Ventricular enddiastolic volume (LVEDV) measured using 2-dimensional echocardiography. The endocardium is traced at end-diastole (frame before mitral valve closure or maximum cavity dimension) in the 2- and 4-chamber views to calculate volumes. Population: All available data has been reported.
  mL
    number analyzed (Participants) | 451
    (all) | 160.26 (75.31)
Serum Creatinine [Mean (Standard Deviation); unit: mg/dl] — Population: All available data has been reported.
  mg/dl
    number analyzed (Participants) | 498
    (all) | 1.71 (1.54)
Brain Natriuretic Peptide (BNP) [Mean (Standard Deviation); unit: pg/mL] — Population: All available data has been reported
  pg/mL
    number analyzed (Participants) | 407
    (all) | 567.11 (766.67)
N-terminal Prohormone of Brain Natriuretic Peptide (NT-proBNP Levels) [Mean (Standard Deviation); unit: Pg/mL] — Population: All available data has been reported
  Pg/mL
    number analyzed (Participants) | 173
    (all) | 6808.17 (17329.44)

OUTCOME MEASURES:

1. Primary Outcome: Single Leaflet Device Attachment (SLDA) Rate
Description: SLDA is defined as the attachment of one mitral leaflet to the MitraClip® Device
Time Frame: up to 30 Days
Population: All subjects with available data were included for analysis.
Measure: Number; unit: percentage of SLDAs
Arm/Group | MitraClip NT System
Number analyzed (Participants) | 497
percentage of SLDAs | 1.21

2. Primary Outcome: No of Participants With Acute Procedural Success (APS)
Description: APS is defined as resulting MR reduction to ≤ 2+ per echocardiographic assessment.
  Mitral regurgitation severity is determined based on the American Society of Echocardiography (ASE) Recommendations for Evaluation of The Severity of Native Valvular Regurgitation with Two-Dimensional and Doppler Echocardiography. MR severity grade was assessed by the core lab using the transthoracic echocardiogram (TTE) at baseline, discharge and subsequent follow-up visits. The severity of MR is determined by the amount of blood being pushed back into the left atrium when it should be circulating through the left ventricle with each heart beat. MR severity is typically classified as mild (grade 1+), moderate (grade 2+), moderate to severe (grade 3+) or severe (grade 4+).
Time Frame: up to 7 days (Discharge visit) from Procedure date
Population: All subjects with available data were used for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | MitraClip NT System
Number analyzed (Participants) | 496
Participants | 452

ADVERSE EVENTS:
Time Frame: This section includes Adverse events reported through 3 years. Subject follow-up is complete.
Arm/Group | MitraClip NT System
All-Cause Mortality (participants affected / at risk) | 163/500
Serious Adverse Events (participants affected / at risk) | 322/500
Other Adverse Events (participants affected / at risk) | 25/500
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MitraClip NT System (N=500)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 (1)
Haemolytic Anaemia (Blood and lymphatic system disorders) | 1 (1)
Hypochromic Anaemia (Blood and lymphatic system disorders) | 1 (1)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 (1)
Angina Pectoris (Cardiac disorders) | 1 (1)
Angina Unstable (Cardiac disorders) | 1 (1)
Aortic Valve Stenosis (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 3 (3)
Atrial Fibrillation (Cardiac disorders) | 12 (17)
Atrial Tachycardia (Cardiac disorders) | 2 (2)
Atrial Thrombosis (Cardiac disorders) | 1 (1)
Atrioventricular Block Complete (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 3 (3)
Cardiac Failure (Cardiac disorders) | 142 (241)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1)
Cardiac Tamponade (Cardiac disorders) | 3 (3)
Cardiogenic Shock (Cardiac disorders) | 2 (2)
Chordae Tendinae Rupture (Cardiac disorders) | 1 (1)
Coronary Artery Stenosis (Cardiac disorders) | 1 (1)
Intracardiac Thrombus (Cardiac disorders) | 1 (1)
Mitral Valve Incompetence (Cardiac disorders) | 24 (24)
Mitral Valve Prolapse (Cardiac disorders) | 9 (9)
Mitral Valve Stenosis (Cardiac disorders) | 1 (1)
Myocardial Ischaemia (Cardiac disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 5 (5)
Sinus Arrest (Cardiac disorders) | 1 (1)
Tricuspid Valve Incompetence (Cardiac disorders) | 1 (1)
Ventricular Fibrillation (Cardiac disorders) | 4 (5)
Ventricular Tachycardia (Cardiac disorders) | 13 (17)
Atrial Septal Defect (Congenital, familial and genetic disorders) | 8 (8)
Vertigo Positional (Ear and labyrinth disorders) | 1 (1)
Basedow's Disease (Endocrine disorders) | 1 (1)
Cataract (Eye disorders) | 4 (4)
Glaucoma (Eye disorders) | 2 (2)
Breath Odour (Gastrointestinal disorders) | 1 (1)
Gastric Ulcer (Gastrointestinal disorders) | 2 (2)
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2)
Intestinal Ischaemia (Gastrointestinal disorders) | 2 (2)
Oesophageal Perforation (Gastrointestinal disorders) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 29 (29)
Multi-Organ Failure (General disorders) | 1 (1)
Sudden Cardiac Death (General disorders) | 1 (1)
Bile Duct Stone (Hepatobiliary disorders) | 3 (3)
Cholangitis Acute (Hepatobiliary disorders) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 1 (1)
Appendicitis Perforated (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1)
Endocarditis (Infections and infestations) | 3 (3)
Herpes Zoster (Infections and infestations) | 2 (2)
Infection (Infections and infestations) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 20 (21)
Pneumonia Bacterial (Infections and infestations) | 1 (1)
Psoas Abscess (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 8 (8)
Septic Shock (Infections and infestations) | 3 (3)
Staphylococcal Infection (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Compression Fracture (Injury, poisoning and procedural complications) | 4 (4)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 5 (5)
Fracture (Injury, poisoning and procedural complications) | 3 (3)
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1)
Pelvic Fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal Cord Injury Cervical (Injury, poisoning and procedural complications) | 1 (1)
Subdural Haematoma (Injury, poisoning and procedural complications) | 3 (3)
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1)
Vascular Access Complication (Injury, poisoning and procedural complications) | 1 (1)
Venous Injury (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 6 (6)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Gallbladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3)
Hepatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Haemorrhagic Stroke (Nervous system disorders) | 6 (6)
Hepatic Encephalopathy (Nervous system disorders) | 1 (1)
Hypoglycaemic Coma (Nervous system disorders) | 1 (1)
Intracranial Aneurysm (Nervous system disorders) | 1 (1)
Ischaemic Stroke (Nervous system disorders) | 9 (10)
Depression (Psychiatric disorders) | 2 (2)
Azotaemia (Renal and urinary disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 25 (25)
Renal Failure Acute (Renal and urinary disorders) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 13 (14)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Henoch-Schonlein Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Cardiac Pacemaker Replacement (Surgical and medical procedures) | 1 (1)
Haemodialysis (Surgical and medical procedures) | 1 (1)
Aortic Dissection (Vascular disorders) | 2 (2)
Arteriosclerosis (Vascular disorders) | 2 (2)
Embolism (Vascular disorders) | 3 (3)
Haemorrhage (Vascular disorders) | 19 (19)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 2 (3)
Peripheral Embolism (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 2 (2)
Congestive Cardiomyopathy (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 2 (2)
Sick Sinus Syndrome (Cardiac disorders) | 3 (3)
Ventricular Dyssynchrony (Cardiac disorders) | 1 (1)
Duodenal Ulcer (Gastrointestinal disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Perforation (Gastrointestinal disorders) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (4)
Device Battery Issue (General disorders) | 1 (1)
Device Deployment Issue (General disorders) | 3 (3)
Device Power Source Issue (General disorders) | 1 (1)
Hernia (General disorders) | 1 (1)
Implant Site Haemorrhage (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Sudden Death (General disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Device Related Sepsis (Infections and infestations) | 1 (1)
Tooth Abscess (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Heat Stroke (Injury, poisoning and procedural complications) | 1 (1)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 (1)
Tendon Rupture (Injury, poisoning and procedural complications) | 1 (1)
International Normalised Ratio Increased (Investigations) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 2 (2)
Carcinoma In Situ Of Eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastrointestinal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases To Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Cerebrovascular Accident (Nervous system disorders) | 1 (1)
Encephalitis (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 3 (3)
Uterine Prolapse (Reproductive system and breast disorders) | 1 (2)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Central Venous Catheterisation (Surgical and medical procedures) | 1 (1)
Implantable Defibrillator Insertion (Surgical and medical procedures) | 1 (1)
Leg Amputation (Surgical and medical procedures) | 1 (1)
Aortic Stenosis (Vascular disorders) | 1 (1)
Aortic Valve Disease (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MitraClip NT System (N=500)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac Failure (Cardiac disorders) | 2 (2)
Chordae Tendinae Rupture (Cardiac disorders) | 1 (1)
Mitral Valve Incompetence (Cardiac disorders) | 3 (3)
Mitral Valve Prolapse (Cardiac disorders) | 2 (2)
Mitral Valve Stenosis (Cardiac disorders) | 4 (5)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 1 (1)
Atrial Septal Defect (Congenital, familial and genetic disorders) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Peripheral Artery Aneurysm (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Device Deployment Issue (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-01-04): https://cdn.clinicaltrials.gov/large-docs/92/NCT03500692/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/92/NCT03500692/SAP_001.pdf